CLINICAL TRIAL: NCT05574751
Title: Laparoscopic Transabdominal Preperitoneal Surgical Repair of Inguinal Hernia Using Sutured Repair Versus Tacker Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damanhour Teaching Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DTH: 22002
Record Dates: First submitted 2022-10-07; First posted 2022-10-12 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-01

CONDITIONS: Inguinal Hernia Unilateral
Keywords: Inguinal hernia; Mesh fixation; Titanium tacker
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Titanium tacker group (n=30) (Active Comparator): Group A
  Interventions: Other: Titanium tacker
- Polypropylene group (n=30) (Active Comparator): Group B
  Interventions: Other: Polypropylene 0

INTERVENTIONS:
Other: Titanium tacker — Mesh fixation with Titanium tacker
  Arms: Titanium tacker group (n=30)
Other: Polypropylene 0 — Mesh was sutured and fixed with polypropylene 0
  Arms: Polypropylene group (n=30)

SUMMARY:
Background: Mesh fixation is a critical step in laparoscopic Transabdominal Preperitoneal (TAPP) hernia repair because fixation is a significant step to prevent the hazard of mesh migration, but is supposed to be associated with a higher risk of acute and chronic pain compared with non-fixation. Fixation is more expensive than non-fixation.

Objective: To compare the efficiency of mesh fixation in laparoscopic TAPP surgical repair of inguinal hernia using sutured repair versus tacker use.

Patients and Methods: This prospective randomized comparative study was carried out on 60 patients who presented with a unilateral inguinal hernia and were assigned to laparoscopic TAPP hernia repair. Patients were randomly allocated into two equal groups (30 patients each); in group A, the mesh was fixed with a Titanium tacker, and in group B, the mesh was sutured and fixed with polypropylene 0.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 21 years
* American Society of Anesthesiologists (ASA) physical status ≤ II
* Patients with body mass index (BMI) of 25 to 35 kg/m²
* Unilateral inguinal hernia

Exclusion Criteria:

* Age < 21 years
* ASA physical status > II
* Patients with body mass index (BMI) > 35 kg/m²
* Pregnant women
* Bilateral inguinal hernia
* Large inguinoscrotal hernia
* Incarcerated hernia
* Recurrent hernia
* Strangulated hernia
* Prostatic diseases
* History of; Convulsions, Cerebrovascular accident, Previous neurological diseases
* Dysrhythmia
* Hypertension
* Ischemic heart disease
* Hyperthyroidism
* Liver or Renal impairment
* Alcohol or drug abuse

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Median and Range of Numeric Pain Rating Scale (NPRS) score [(median (range)] | 7 days after the end of the operation
  NPRS measures the severity of postoperative pain, it is a 11 point scale from 0-10; where 0=No pain and 10=Worst possible pain (2h, 6h, 12h, 24h, 48h, 72h, and 7 days)
Mean and Standard deviation of Numeric Pain Rating Scale (NPRS) score (mean±SD) | 7 days after the end of the operation
  NPRS measures the severity of postoperative pain, it is a 11 point scale from 0-10; where 0=No pain and 10=Worst possible pain (2h, 6h, 12h, 24h, 48h, 72h, and 7 days)

SECONDARY OUTCOMES:
Mean and Standard deviation of Operative duration (minutes) (mean±SD) | 2 minutes after the end of the operation
  Time from skin incision till skin closure
Mean and Standard deviation of Length of hospital stay (hours) (mean±SD) | 24 hours after the end of the operation
  Time from hospital admission till discharge
Number of participants and Rate of Intraoperative complications | 2 minutes after the end of the operation
  Number of participants and Rate of: Bowel injury, Injury to inferior epigastric artery, Injury to major vessels, Bleeding of venous plexus around pubic bone, Injury to vas deferens, Bladder injury.
Number of participants and Rate of Postoperative complications | 1 year after the end of the operation
  Number of participants and Rate of: Cord edema, Seroma, Port-site infection, Inguinal anesthesia/hyperthesia, Chronic pain, Recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Shaat, MD, Principal Investigator — Damanhour Teaching Hospital
Locations (1):
- Damanhour Teaching Hospital, Damanhūr, El-Beheira, Egypt